**PRINCIPAL INVESTIGATOR:** Anish Thomas, M.D.

STUDY TITLE: A Phase I/II Trial of Topotecan with VX-970 (M6620), an

ATR Kinase Inhibitor in Small Cell Cancers

STUDY SITE: NIH Clinical Center

Cohort: Affected Patient

Consent Version: 06/12/2020

#### WHO DO YOU CONTACT ABOUT THIS STUDY?

# **Principal Investigator:**

Thomas Anish, MD Phone: 240-760-7343

Email: anish.thomas@nih.gov

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). Members of the study team will talk with you about the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). Take the time needed to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers. Taking part in research at the NIH is your choice.

If the individual being asked to participate in this research study is not able to give consent for themselves, you, as the Legally Authorized Representative, will be their decision-maker and you are being asked to give permission for this person to be in this study. For the remainder of this document, the term "you" refers to you as the decision-maker and/or the individual being asked to participate in this research.

#### IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### WHY IS THIS STUDY BEING DONE?

Patients with cancer may stop responding to chemotherapy over time. Most patients who stop responding to their initial chemotherapy are then treated with a different type of chemotherapy.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/12/2020


Most chemotherapies work by damaging the DNA in the cancer cells, causing those cells to die and the tumor to shrink.

However, chemotherapy alone may not be effective at causing cancer cell death. Research shows that some tumor cells can be less affected by chemotherapy because they have ways to repair the damaged DNA. One of the pathways to repair DNA involves a protein called ataxia telangiectasia and Rad3-related (ATR). Our research in the laboratory suggests that giving chemotherapy along with another drug which restricts ATR will block that DNA repair process, causing the tumor cells to die.

The purpose of this study is to examine whether using chemotherapy together with a drug which inhibits ATR will lead to an increase in the death of cancer cells, and therefore a better response to treatment in cancer patients. For this trial, we are using the chemotherapy drug, topotecan, with a drug called M6620 which inhibits ATR. M6620 is an investigational agent, meaning that it has not been approved by the US FDA for the treatment of your cancer. Topotecan is approved by the FDA for use in small cell lung cancer, ovarian cancer and in cancers of the cervix. Although not approved for the treatment of any other types of cancer, small studies have shown that topotecan may have antitumor effect in a number of other cancers, including neuroendocrine tumors and non-small cell lung cancer.

This study is divided into two parts, Phase I and Phase II. The Phase I portion of the study is being done to test the safety of the combination of M6620 and topotecan, and to determine the highest doses of these two drugs that can be given in combination safely in patients with a variety of cancers. During Phase II, this study will analyze how effective this drug combination is in treating small cell cancers.

## WHY ARE YOU BEING ASKED TO TAKE PART IN THIS STUDY?

You have been asked to take part in this study because you have been diagnosed with SCLC or an extra-pulmonary small cell carcinoma. Small cell cancers can arise in the lungs and less commonly in other parts of the body. These tumors share many similarities including their fast growth and limited response to treatment when it comes back after initial chemotherapy.

## HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

Up to 70 people will take part in this study; this includes Phase I and II.

## DESCRIPTION OF RESEARCH STUDY

#### Before you begin the study

Before you begin this study, you will have several exams and tests to make sure you are eligible for this study. Most of the tests needed would be part of your routine medical care for your cancer and are performed under a separate consent. They include blood tests, physical examination, an EKG and CT scans. If you are a woman who can become pregnant, you will also have a pregnancy

If it is determined that you are eligible for the study and you chose to sign the consent, you will be enrolled onto the study.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

ÍRB NUMBER: 15C0150 Version Date: 06/12/2020 IRB APPROVAL DATE: 06/22/2020


# **During the study**

You will receive topotecan on days 1 to 5 and M6620 on day 5 or days 2 and 5 (depending on the drug dose, see paragraph below and study chart) of each 21-day cycle. You will continue to receive treatment until your disease no longer responds or you are no longer able to tolerate the drug. You will receive both medications intravenously (IV). Topotecan will be administered for approximately 30 minutes and M6620 for approximately 60 minutes.

Subjects will initially be enrolled on the study in groups of 3 or 6. The first group will take topotecan and M6620 at the starting pre-planned dose. If none or only one of the subject experiences intolerable side effects, the next group will be enrolled at the next highest dose. This will continue until more than one person in a group has intolerable side effects or until the highest pre-planned dose has been reached. The maximum safe dose is set at the highest dose in which no more than one of six participants experienced an intolerable side effect.

Once the maximum safe dose is determined, in the second part of the study (phase 2), up to 25 subjects will be enrolled at that dose to evaluate the anti-cancer activity of topotecan with M6620 in small cell lung cancer.

If you experience side effects (described later in this consent) when taking topotecan and/or M6620, the dosage of these drugs may be adjusted to reduce the severity of your side effects. Also, subsequent doses may be delayed until you have time to recover. If the side effects are too severe, the doctor may decide to stop all further doses of topotecan and/or M6620.

During the first cycle, the health care provider will monitor you weekly. After the first cycle, these check-ups will be performed every three weeks. If your doctor believes that it is necessary, based on your symptoms, the physical exam will be performed more often than indicated. Please see the study chart for the schedule of the tests.

#### **Research Studies**

An important part of the research is to determine how your body and tumor responds to the combination of drugs. To understand this, we will collect your blood, hair samples and tumor at different time points. Single hairs will be plucked from the scalp with forceps. Plucked hairs from eyebrows will be collected only if we cannot get hair from your scalp.

Biopsies will be optional. If you agree to have the biopsies, these will be performed before you start treatment, on day 3 of cycle one, and if you stop responding to the drug or your disease worsens. If you are participating in Phase I and are receiving the lowest dose of topotecan and M6620, you will have only one biopsy performed (on day 3 of treatment). You will be asked to sign a separate consent for the biopsy at the time of the procedure.

We will be using the biopsies and blood samples to look at the genes (pieces of DNA) that are present in tumor cells and in blood cells. This information may help us understand why some patients respond to certain treatments better than the others. In the course of examining your DNA, it is possible that we could identify possible changes in genes that are not the target of our investigation, but which are associated with diseases. These are called incidental or secondary findings. The analyses that we perform in our laboratory are for research purposes only; they are not nearly as sensitive as the tests that are performed in a laboratory that is certified to perform genetic testing. Changes that we observe unrelated to our research may or may not be valid.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/12/2020 Page **3** of **17**  Therefore, we do not plan to inform you of the results of testing on your specimens that is performed in our research lab. However, in the unlikely event that we discover a finding that is believed to be clinically important based on medical standards at the time we first analyze your results, we will contact you. This could be many years in the future. We will ask you to have an additional tube of blood drawn to verify the findings we have seen in our lab. If the results are verified, you will be re-contacted and offered a referral to a genetic healthcare provider to discuss the results.

Please see the section discussing the risks that you might experience other than the drug side effects for the implications of receiving genetic information.

We may also collect your blood on the first two days of the first cycle in order to see how quickly study medications are metabolized in your blood. These are called pharmacokinetic studies. If you are scheduled to participate in these research studies, on day 1 of cycle 1, we will collect your blood before you start topotecan infusion, at the end of infusion, 30 minutes after the end of infusion and then 1, 2, 4, 8 and 24 hours after the end of infusion. On day 2 of cycle 1, we will collect your blood before you start M6620 infusion, at the end of infusion, 30 minutes after the end of infusion and then 1, 4, 8, 24 and 48 hours after the end of infusion. On both of those days, you will have to be admitted to a hospital overnight.

# When you are finished taking the drugs (treatment)

In the case that you have to stop receiving treatment, you will have a clinic visit approximately 4 weeks after you discontinue taking the study drugs, in which the health care provider will perform a physical exam and blood will be drawn. You will then receive follow-up phone calls from the study team every three months.

## STUDY CHART

| Day | What to do and what will happen to you |
|---|---|
| Before<br>starting | The research team's health care provider will go over your medical his and will perform a physical exam. |
| | Blood samples will be collected. |
| | An echocardiogram and CT scan will be performed. |
| | You will have a pregnancy test if you are a woman who can become pregnant. |
| | An optional tumor biopsy will be performed, depending on to which group you are assigned, and if you agree. |

## Cycle 1

| Day 1 | The research team's health care provider will perform a physical exam. |
|---|---|
| | * Blood samples will be collected. |
| You will have a pregnancy test if you are a woman who can become p | |
| | Hair samples will be collected. |

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


| | You will receive the first dose of topotecan IV. |
|---|---|
| Day 2 | You will receive the second dose of topotecan and the first dose of M6620 (depending on to which group you have been assigned) IV. |
| | If you are receiving the first dose of M6620, you will undergo an ECG before and after the M6620 infusion. |
| | * Blood and hair samples will be taken. |
| Day 3 | You will receive third dose of topotecan IV. |
| | Blood and hair samples will be taken. |
| | An optional biopsy will be performed if you agree. |
| Day 4 | You will receive the fourth dose of topotecan IV. |
| Day 5 | The research team's health care provider will perform a physical exam. |
| | You will receive the fifth dose of topotecan and the first or second dose of M6620, depending on to which group you have been assigned, IV. |
| | If you are receiving the first dose of M6620, you will undergo an ECG before and after the M6620 infusion. |
| | Blood samples may be collected. |
| Day 8 | Blood samples will be collected for assessing blood counts, liver and kidney functions |
| Day 15 | Blood samples will be collected for assessing blood counts, liver and kidney functions |

<sup>\*</sup> If you are scheduled to participate in these research studies, you will have to be admitted to a hospital overnight on this day in order to collect blood for pharmacokinetic studies.

# Cycle 2 and beyond

| Day 1 | The research team's health care provider will perform a physical exam. Blood samples will be collected. You will have a pregnancy test if you are a woman who can become pregnant. You will receive topotecan IV. |
|---|---|
| Day 2 | You will receive topotecan IV. You will receive M6620 depending on the dose group to which you were assigned. |
| Day 3 | You will receive topotecan IV. |

**PATIENT IDENTIFICATION** 

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/12/2020 Page **5** of **17**  ÍRB NUMBER: 15C0150 IRB APPROVAL DATE: 06/22/2020

| Day 4 | You will receive topotecan IV. |
|---|---|
| Day 5 | The research team's health care provider will perform a physical exam. You will receive topotecan and M6620 IV. |
| Day 8 | Blood samples will be collected for assessing blood counts, liver and kidney functions (Cycle 2 only) |
| Day 15 | Blood samples will be collected for assessing blood counts, liver and kidney functions (Cycle 2 only) |
| Day 21 | A CT scan will be performed after every 2 cycles |
| Off Treatment | |
| | The research team's health care provider will go over your medical history and will perform a physical exam. |
| | Blood samples will be collected. |
| | An optional tumor biopsy will be performed, depending on to which group you are assigned, and if you agree. |
| | You will receive follow-up phone calls every 3 months |

<u>Note:</u> At each study visit, you will be able to report any side effects that you have experienced to the research team.

## **BIRTH CONTROL**

If you are a woman who is breast feeding or pregnant, you may not take part in the study because we don't know how this medicine would affect your baby or your unborn child. If you are a woman who can become pregnant, or are the partner of a woman who can become pregnant, you will need to practice an effective form of birth control before starting study treatment and during study treatment, and for 6 months after you finish study treatment. If you think that you or your partner is pregnant, you should tell your study doctor or nurse at once.

Effective forms of birth control include:

- abstinence
- intrauterine device (IUD)
- hormonal [birth control pills, injections, or implants]
- tubal ligation
- vasectomy

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


IRB NUMBER: 15C0150
IRB APPROVAL DATE: 06/22/2020

## RISKS OR DISCOMFORTS OF PARTICIPATION

#### From M6620

M6620 has been studied in multiple doses either by itself or in combination with a chemotherapeutic agent in subjects with advanced cancer. M6620, by itself or with a chemotherapeutic agent, can have some unwanted effects.

M6620 may cause an infusion reaction. In some subjects, this is a reaction limited to the body site where the drug is being infused, for example swelling, itching, and/or redness around the site. In some subjects, the reaction is a whole-body reaction, for example flushing and/or redness everywhere, and/or nausea, headache or other symptoms.

M6620 infrequently (<5% of subjects) causes a serious infusion reaction, with symptoms including flushing, shortness of breath, low blood pressure, feeling of faintness, sweating and abdominal discomfort. These symptoms have resolved after stopping the infusion and treating the reaction with other intravenous (IV) medications. The Study doctor may treat this with medications, and try to decrease the chances of these side effects occurring in the future by giving you medication to avoid these symptoms in advance of the infusion or by slowing down the rate of infusion.

Intravenous (IV) infusion of M6620 may cause local irritation, redness, tenderness, or rash at the injection site. Many of these local side effects go away after the infusion is stopped or standard measures are applied to treat the symptoms including removing and replacing the catheter or slowing the rate of infusion.

Risks due to M6620 alone:

- Nausea 32%
- Vomiting 12%
- Infusion site reactions (occur at the body site where the drug is infused) 9%
- Systemic infusion reactions (affect the whole body) 17%

Risks when M6620 is given with chemotherapy:

- Nausea 54%
- Vomiting 33%
- Infusion site reactions (occur at the body site where the drug is being infused) 10%
- Systemic infusion reactions (affect the whole body) 15%

Additional risks of M6620 given in combination with carboplatin:

- Anemia 52%
- Low neutrophils (a type of immune cells that are involved in fighting infections) 45%
- Low platelets (cells that play a role in stopping bleeding) 38%

In addition, the following very common adverse events were observed in at least 15% of subjects receiving M6620 monotherapy. There is not enough experience in M6620 whether these truly are side effects.

- Diarrhea 15%
- Fatigue (feeling tired) 20%

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


There is a possibility that M6620 may make you more sensitive to sunlight. You should limit your exposure to the sun, including exposure to sunlamps and tanning beds. Use of sun block and wearing long sleeved clothing and sunglasses is recommended.

There may be other side effects that we cannot predict, but your Study doctors have taken steps to minimize the risks. During this Study, your doctor will ask you about any symptoms you may experience. In addition, you will be monitored for side effects that you may not have symptoms from but are seen through lab testing, including, abnormal liver tests and abnormal blood counts including platelets, white blood cells, and red blood cells. Many side effects go away on their own with time or after using other medications to treat them.

There may be risks and side effects from the M6620 that are not yet known. You should call your study doctor if you think you are having any of the problems listed above or even if you are having problems that are not on the list.

In addition, as with any medication including over-the-counter medications, there is a small but significant risk of allergic reactions that, if severe, can be fatal. These types of reactions can start shortly after taking a medication and may appear in the form of itching or redness of the skin, swelling of the face, lips, tongue, throat, or difficulty breathing which may be severe in some cases. If you experience any of these reactions, you must let the Study doctor know immediately, and, if you are not in the hospital at the time you are having the reaction, you should call 911 or go to the closest Emergency Department for treatment. If this happens, you should tell the treating physician that you are in a Study. You will be given a wallet card to carry with you which will have information about the Study you are in.

# From topotecan

# Likely, some may be serious (experienced by more than 20% of persons taking the drug)

- Anemia which may require a blood transfusion
- Low white blood cell counts
- Constipation, diarrhea, nausea, vomiting
- Fever
- Pain
- Bruising, bleeding
- Infection, especially when white blood cell count is low
- Tiredness
- Shortness of breath

# Less likely, some may be serious (experienced by between 3 and up to 20% of persons taking the drug)

- Sores in mouth which may cause difficulty swallowing
- Headache
- Cough
- Scarring of the lungs

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

IRB APPROVAL DATE: 06/22/2020

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/12/2020 IRB NUMBER: 15C0150


## Rare but Serious (experienced by 3% of fewer of persons taking the drug)

- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Low white blood cell counts which may result in life-threatening infections

Note: Some of the side effects associated with these drugs could potentially lead to death.

# Risks you might experience other than the drug side effects

## **Biopsy Risk**

Risks associated with the biopsies are pain and bleeding at the biopsy site. Sometimes a CT scan may be needed to identify the right tumor to biopsy.

#### **Radiation Risk**

During your participation in this research study, you will be exposed to radiation from 3 CT guided biopsies and 9 CT scans. The amount of radiation exposure you will receive from these procedures is equal to approximately 12.3 rem. A rem is a unit of absorbed radiation.

Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. The average person in the United States receives a radiation exposure of 0.3 rem per year from these sources. This type of radiation is called "background radiation." This study will expose you to more radiation than you get from everyday background radiation. No one knows for sure whether exposure to these low amounts of radiation is harmful to your body.

The CT scans that you get in this study will expose you to roughly the same amount of radiation as 41 years' worth of background radiation. Being exposed to too much radiation can cause harmful side effects such as an increase in the risk of cancer. The risk depends on how much radiation you are exposed to. Please be aware that about 40 out of 100 people (40%) will get cancer during their lifetime, and 20 out of 100 (20%) will die from cancer. The risk of getting cancer from the radiation exposure in this study is 1.2 out of 100 (1%) and of getting a fatal cancer is 0.6 out of 100 (0.5%).

## Radiation Exposure in People Capable of Becoming Pregnant

You may not participate in this study if you are pregnant. If you are able to become pregnant, we will perform a pregnancy test before exposing you to radiation. You must tell us if you may have become pregnant within the previous 14 days because the pregnancy test is unreliable during that time.

#### CT contrast risk

Itching, hives (small bumps on the skin) or headaches are possible risks associated with contrast agents that may be used during CT imaging. Symptoms of a more serious allergic reaction include shortness of breath and swelling of the throat or other parts of the body. Very rarely, the contrast agents used in CT can cause kidney problems for certain patients, such as those with impaired kidney function.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

ÍRB NUMBER: 15C0150 Version Date: 06/12/2020 IRB APPROVAL DATE: 06/22/2020


## **Blood Draw Risk**

Risks associated with blood draw include pain and bruising, lightheadedness, and rarely, fainting

# **Hair Sample Collection Risk**

You may experience pain associated with hair collection.

# Psychological or Social Risks Associated with Loss of Privacy in Genetic Research

As part of the research study, it is possible that you could learn that you have genetic risks for another disease or disability. This may be upsetting and, depending on what you learn, might create a need to make challenging decisions about how to respond.

Although your genomic information is unique to you, you share some genomic similarities with your children, parents, brothers, sisters, and other blood relatives. Therefore, learning your research results could mean something about your family members and might cause you or your family distress. Before joining the study, it may be beneficial to talk with your family members about whether and how they want you to share your results with them.

# Privacy Risks Associated with Return of Incidental or Secondary Findings

Although your genetic information is unique to you, you do share some genetic information with your children, parents, brothers, sisters, and other blood relatives. Consequently, it may be possible that genetic information from them could be used to help identify you. Similarly, it may be possible that genetic information from you could be used to help identify them. Patterns of genetic variation also can be used by law enforcement agencies to identify a person or his/her blood relatives.

## Protections against misuse of genetic information

This study involves genetic testing on samples. Some genetic information can help predict future health problems of you and your family and this information might be of interest to your employers or insurers. The Genetic Information Nondiscrimination Act (GINA) is a federal law that prohibits plans and health insurers from requesting genetic information or using genetic information. It also prohibits employment discrimination based on your health information. However, GINA does not address discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA also does not protect you against discrimination based on an already-diagnosed condition or disease that has a genetic component.

## POTENTIAL BENEFITS OF PARTICIPATION

## Are there benefits to taking part in this study?

The aim of this study is to see if this experimental combination treatment will cause your tumors to shrink. We do not know if you will receive personal, medical benefit from taking part in this study. These potential benefits could include shrinking of your tumor or lessening of your symptoms, such as pain, that are caused by the cancer. Because there is not much information about the effect of this drug combination on your cancer, we do not know if you will benefit from taking part in this study, although the knowledge gained from this study may help others in the future who have cancer

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


## ALTERNATIVE APPROACHES OR TREATMENTS

#### WHAT OTHER CHOICES DO I HAVE IF I DO NOT TAKE PART IN THIS STUDY?

Instead of being in this study, you have these options:

- Getting treatment or care for your cancer without being in a study
- Taking part in another study
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly. Instead, it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Please talk to your doctor about these and other options.

## STOPPING THERAPY

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease is no longer responding to treatment. Your study doctor will discuss this in detail with you.
- if you have side effects from the treatment that your doctor thinks are too severe
- if new information shows that another treatment would be better for you

In this case, you will be informed of the reason therapy is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to the sponsor of the pharmaceutical company providing the drug and their designated representatives. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases cannot be recalled and destroyed.

# CERTIFICATE OF CONFIDENTIALITY

To help us protect your privacy, we have obtained a Certificate of Confidentiality. The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

You should also know that there are several circumstances in which the Certificate does not provide coverage. These include when information:

PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


ÍRB NUMBER: 15C0150  IRB APPROVAL DATE: 06/22/2020

- will be used for auditing or program evaluation internally by the NIH; or
- must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA).
- is necessary for your medical treatment and you have consented to this disclosure;
- is for other research.

In addition, identifiable, sensitive information protected by this Certificate cannot be admissible as evidence or used for any purpose in any action, suit, or proceeding without your consent.

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

The Certificate of Confidentiality will not protect against the required reporting by hospital staff of information on suspected child abuse, reportable communicable diseases, and/or possible threat of harm to self or others.

# **CONFLICT OF INTEREST**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a Protocol Review Guide. You may ask your research team for a copy of the Protocol Review Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines but they do not need to report their personal finances to the NIH.

Members of the research team working on this study may have up to \$15,000 of stock in the companies that make products used in this study. This is allowed under federal rules and is not a conflict of interest.

The National Institutes of Health and the research team for this study are using a drug (M6620) developed by EMD Serono through a joint study with your researchers and the company. The company also provides financial support for this study.

## USE OF SPECIMENS AND DATA FOR FUTURE RESEARCH

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

We would like to keep some of your specimens and data that we collect for future research and share them with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your specimens and data will be for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and/or data. Then any specimens that have not already been used or shared will be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

# **Genomic Data Sharing**

As part of this research study, we will put your genomic data in a large database for broad sharing with the research community. These databases are commonly called data repositories. The information in this database will include but is not limited to genetic information, race and ethnicity, and sex. If your individual data are placed in one of these repositories, they will be labeled with a code and not with your name or other information that could be used to easily identify you, and only qualified researchers will be able to access them. These researchers must receive prior approval from individuals or committees with authority to determine whether these researchers can access the data.

Summary information about all of the participants included in this study (including you) is being placed in a database and will be available through open access. That means that researchers and non-researchers will be able to access summary information about all the participants included in the study, or summary information combined from multiple studies, without applying for permission. The risk of anyone identifying you with this information is very low.

NIH policies require that genomic data be placed in a repository for sharing. Therefore, we cannot offer you a choice of whether your data will be shared. If you do not wish to have your data placed in a repository, you should not enroll in this study.

## COMPENSATION, REIMBURSEMENT, AND PAYMENT

## Will you receive compensation for participation in the study?

Some NIH Clinical Center studies offer compensation for participation in research. The amount of compensation, if any, is guided by NIH policies and guidelines.

You will not receive compensation for participation in this study.

## Will you receive reimbursement or direct payment by NIH as part of your participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

On this study, the NCI will cover the cost for some of your expenses. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. The amount and form of these payments are determined by the NCI Travel and Lodging Reimbursement Policy. You will be given a summary of the policy which provides more information.

## Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


- CONSENT TO PARTICIPATE IN AN NIH CLINICAL RESEARCH STUDY
- If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

## CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database. Your test results will be identified by a unique code and the list that links the code to your name will be kept separate from your sample and health information. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you.

# Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor (Center for Cancer Research) or their agent(s)
- Qualified representatives from EMD Serono, the pharmaceutical company who produces M6620.

The researchers conducting this study and the NIH follow applicable laws and policies to keep your identifying information private to the extent possible. However, there is always a chance that, despite our best efforts, your identity and/or information about your participation in this research may be inadvertently released or improperly accessed by unauthorized persons.

In most cases, the NIH will not release any identifiable information collected about you without your written permission. However, your information may be shared as described in the section of this document on sharing of specimens and data, and as further outlined in the following sections.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

## **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical records we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your medical record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

## POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


## PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Anish Thomas MD, <a href="mailto:anish.thomas@nih.gov">anish.thomas@nih.gov</a>, 240-760-7343. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

## **CONSENT DOCUMENT**

Please keep a copy of this document in case you want to read it again.

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/12/2020 Page **16** of **17** 

| Signature of Research Participant | Print Name of Research Participant | Date |
|---|---|---|
| about this study and have been given to make research decisions on behalf o | (LAR) for an Adult Unable to Consent: I have the opportunity to discuss it and to ask questions. If the adult participant unable to consent and have the information in the above consent was described expate in the study. | I am legally authorized the authority to provide |
| Signature of LAR | Print Name of LAR | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | Date |
| Witness to the oral short-form conse | ent process only: | |
| Witness: | | |
| Signature of Witness* | Print Name of Witness | Date |
| *NIH ADMINISTRATIVE SECT INTERPRETER: | ION TO BE COMPLETED REGARDING | THE USE OF AN |
| | I, who speaks English and the participant's prefer<br>at and served as a witness. The investigator obtain | 0 0 |
| | l, who speaks English and the participant's prefer<br>t but <u>did not</u> serve as a witness. The name or ID | code of the person |

CC pre rCR ICF template v. 05.05.2020

File in Section 4: Protocol Consent (1)


IRB NUMBER: 15C0150 IRB APPROVAL DATE: 06/22/2020